Official Title: RADx-UP CDCC Rapid Research Pilot Program: "Culturally-relevant Community Connections (C3) to Increase COVID-19 Testing in the Black/African American Community".

**NCT:** NCT05918952

**IRB Document Date:** 11/20/2023

## RADx-UP CDCC Rapid Research Pilot Program

"Culturally-relevant Community Connections (C3) to increase COVID testing in the Black/African American Community".

You are being asked to take part in this research study because we want to understand testing barriers and facilitators of those who self-identify as black/African American. The purpose of this study is to identify barriers and facilitators to COVID testing among members of the Black/African American community. The expected outcome of this project is to increase COVID testing among Black/African American community. The second aim is to examine the use of culturally relevant edutainment video messaging combined with trusted opinion leaders in the community as a strategy to increase COVID testing.

## WHAT are the NIH and RADx-UP?

The NIH stands for the National Institutes of Health. The NIH supports health research, including the RADx- UP program.

RADx-UP stands for Rapid Acceleration of Diagnostics - Underserved Populations. RADx-UP is a COVID-19 research program.

If you decide to join this study, we will:

- Ask you to take two COVID-19 tests within 48 hrs. You will also be invited to a community conversation on COVID-19 in the black community that will take place once every three months.
- Ask you for basic information such as your name, date of birth, address, contact information, race, ethnicity, gender, language, health insurance status, disability, job, and household information including address history.
- Ask you information about COVID-19, including information about any symptoms (a change in your health) and test results. If you had a positive COVID-19 test, we will ask for information about contact tracing (people who may have come in contact with you while you had COVID-19). We will ask about your medical history and if you have or have not had vaccines and why.
- Ask you information about your health, education, family, home, relationships, and social life, among others.

DUHS IRB

IRB NUMBER: Pro00112394

IRB REFERENCE DATE: 06/28/2023
IRB EXPIRATION DATE: 03/30/2025

- We will ask you to fill out questionnaires, surveys and other forms to collect the information above.
  - Participants have the option to either get Covid testing done onsite, or only watch the edutainment videos and respond to survey questions based only on the edutainment videos.

You will be given a \$5 dollar off coupon towards your service at the designated barbershop or beauty salon collaborating with the research team for consenting to be a part of this study.

There may be direct medical benefit to you. We hope that in the future the information learned from this study will benefit others in the community.

## What WILL YOU DO WITH MY DATA?

Duke was chosen by the NIH to hold the data from all RADx-UP studies. Duke will keep your data securely. This means with extra protection. Researchers will use the data to learn more about COVID-

Duke will build two RADx-UP databases. Databases are systems that hold electronic information.

The first database will only hold data that can easily identify you. These data are called identifiable data. Examples include your name, address, email, and phone number, among others.

- Duke will not share your identifiable data with others.
- Your data will be stored securely. Only study staff approved by a research ethics committee will be able to see your data.

The second database will not hold data that can easily identify you. It will hold all of your other data.

- Your data will be assigned a study code. Your data will only be identified in this database by this study code.
- Your data may be linked with other data using your zip code. This linked data will tell us more about the area where you live.
- We will transfer these data to a secure NIH database. These data will not be able to identify you.
- Other researchers may use these data for future studies.
- We will not ask your permission before sharing these data because they are non-identifiable.

Participation in research involves some loss of privacy. We will do our best to make sure that information about you is kept confidential, but we cannot guarantee total confidentiality.

DUHS IRB

IRB NUMBER: Pro00112394

IRB REFERENCE DATE: 06/28/2023
IRB EXPIRATION DATE: 03/30/2025

Your personal information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding, and regulating the study. We will share only the minimum necessary information to conduct the research.

Your privacy is very important to us. We will take great care to protect your privacy. However, there is always a chance that, even with our best efforts, your identity and/or information collected during this study may be accidentally released or seen by unauthorized persons. Here are a few steps we will take:

- Data will be stored on protected, secure computer systems. We will limit and keep track of who can see these data.
- We will take steps to protect your information from others that should not be able to see it.
- When your data are shared with other researchers, they will not have information that can identify you.

This project has a Certificate of Confidentiality from the United States government. Certificates of Confidentiality protect your privacy by blocking the release of identifiable, sensitive research information to anyone not connected to the research except when you agree, or in a few other specific situations.

"A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time."

If you have questions about your participation, please contact the researcher, Dr. Schenita Randolph by calling contact the researcher contact the researc

If you have questions, concerns, or a complaint about your involvement in a research study or your rights as a research participant, please contact the Duke Institutional Review Board by calling 919-668-5111.

Please be advised that you do not have to take part in this study. Being in this study will not change health care for you or your family member at Duke University Health System or its affiliates. You can guit this study at any time.

Would you like to participate in this study?

If you choose not to take a COVID test, we will collect data on the reason for your decision. If you say yes to testing, we will also collect data. For either route, you will receive a \$5 off coupon.

By proceeding to watch the video, you consent to taking part in this study.

**DUHS IRB** 

IRB NUMBER: Pro00112394

IRB REFERENCE DATE: 06//28//2023
IRB EXPIRATION DATE: 03/30/2025